CLINICAL TRIAL: NCT06262191
Title: An Adjustable Stiffness Orthosis to Maintain Muscle Engagement and Push-off Power in Cerebral Palsy
Brief Title: Testing an Adjustable Ankle Orthosis During Walking in Cerebral Palsy
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Northern Arizona University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2137249
Record Dates: First submitted 2024-01-29; First posted 2024-02-15 (Actual); Results first posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Study group (Experimental): Participants will walk with the new AFO, their own AFOs, and no AFOs.
  Interventions: Device: Differential and adjustable stiffness AFO (DAS-AFO)

INTERVENTIONS:
Device: Differential and adjustable stiffness AFO (DAS-AFO) — Walking with a differential and adjustable stiffness AFO (DAS-AFO)

SUMMARY:
This study seeks to determine how an adjustable stiffness ankle braces affects walking performance and biomechanics in cerebral palsy.

DETAILED DESCRIPTION:
Our first aim is to confirm that the differential and adjustable stiffness (DAS) AFO improves plantarflexor push-off power and range of motion compared to standard (physician prescribed) AFOs during walking in CP.

Our second aim is to confirm that the differential and adjustable stiffness (DAS) AFO improves plantarflexor muscle activity while maintaining improved posture compared to standard AFOs during walking in CP.

Our third aim is to validate the need and usability of real-time stiffness adjustment during play and school activities; obtain feedback from the children, their parents, and orthotists to design the MVP.

ELIGIBILITY:
Inclusion Criteria:

* Age between 8-35 years old, inclusive
* Diagnosis of cerebral palsy (CP)
* Gross motor functional classification score level I, II, or III
* Physician-prescribed AFOs of common design (i.e., rigid molded thermoplastic)
* Ability to walk for 6 minutes on a treadmill
* At least 20° of passive plantar-flexion range of motion
* No concurrent treatment other than those assigned during the study
* No condition other than CP that would affect safe participation
* No surgery within 6 months of participation.

Exclusion Criteria:

-Excessive knee flexion during walking caused by CP

Ages: 8 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 11 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Northern Arizona University, Flagstaff, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Study Group
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Study Group
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.5 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Change in Muscle Activity
Description: Change in integrated soleus electromyography (mV/mV) muscle activity during stance phase of walking.
Time Frame: day 1
Measure: Mean (Standard Deviation); unit: percent change based on mV/mV measures
Arm/Group | Study Group
Number analyzed (Participants) | 11
percent change based on mV/mV measures | -0.09 (0.10)

2. Primary Outcome: Change in Metabolic Cost of Transport
Description: Change in metabolic cost of transport during walking. To calculate the metabolic cost of transport, the standing baseline metabolic rate for each participant and each trial was subtracted from their walking metabolic rate to estimate the net metabolic rate of walking. Next, we normalized the net metabolic rate of walking by each participant's body mass (m) and walking speed to calculate the metabolic cost of transport (J/kg*m), averaged over the last two minutes of each condition.
Time Frame: day 1
Measure: Mean (Standard Deviation); unit: J/kg*m
Arm/Group | Study Group
Number analyzed (Participants) | 10
J/kg*m | 0.57 (1.16)

3. Primary Outcome: Change in Ankle Power
Description: Change in peak ankle power during stance phase measured in w/kg. Ankle kinematics and kinetics were calculated in OpenSim using the collected three-dimensional motion capture and the ground reaction forces. The joint kinematics and ground reaction forces were filtered using a low pass fourth order recursive Butterworth filter with a cut-off frequency of 6 Hz before being used to calculate joint kinetics. The ground reaction forces were collected using two force places associated with the instrumented treadmill (Bertec Corp, Columbus, USA) collected at 1200 Hz. The resultant joint kinetics were then further filtered using the same filtering parameters. Ankle joint power was calculated as the product of the joint moment and joint angular velocity.
Time Frame: 1 day during walking
Measure: Mean (Standard Deviation); unit: w/kg
Arm/Group | Study Group
Number analyzed (Participants) | 11
w/kg | 0.01 (0.61)

ADVERSE EVENTS:
Time Frame: 2 days during the study protocol
Arm/Group | Study Group
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2024-12-18): https://cdn.clinicaltrials.gov/large-docs/91/NCT06262191/Prot_000.pdf
  • Statistical Analysis Plan (2024-12-18): https://cdn.clinicaltrials.gov/large-docs/91/NCT06262191/SAP_001.pdf
  • Informed Consent Form (2024-12-18): https://cdn.clinicaltrials.gov/large-docs/91/NCT06262191/ICF_002.pdf